CLINICAL TRIAL: NCT04867135
Title: Population Pharmacokinetics of Amikacin in Suspected Cases of Neonatal Sepsis: Multicenter Study
Brief Title: Population Pharmacokinetics of Amikacin in Neonates
Status: Completed | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Other Study IDs: 190325002
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2021-04

CONDITIONS: Neonatal Sepsis, Late-Onset
Keywords: Neonatal Sepsis; Amikacin; Population Pharmacokinetic; Neonate
MeSH Terms: conditions — Neonatal Sepsis | interventions — Amikacin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No Sepsis / Sepsis: To compare amikacin PK / PD models of newborns with a confirmed diagnosis of sepsis (clinical or microbiological) and with ruled out sepsis.
  Interventions: Drug: Amikacin Sulfate Injection

INTERVENTIONS:
Drug: Amikacin Sulfate Injection — The dose and frequency of amikacin was defined by each hospital.
  Other Names: Amikacin

SUMMARY:
Aminoglycosides such as Amikacin are routinely used in newborns for the treatment of neonatal sepsis due to gram-negative bacilli. Despite the frequency of this indication, it has not yet been possible to establish definitive dosage schedules that ensure effectiveness and low risk of toxicity, due to the high pharmacokinetic variability observed in this population.

In addition to anthropometric variables, evidence from retrospective studies suggests that sepsis could be capable of significantly modifying the pharmacokinetics of aminoglycosides in neonates, but the investigators suggest conducting prospective studies of higher methodological quality to verify this hypothesis.

Due to the lack of pharmacokinetic and pharmacodynamic (PK / PD) studies of Amikacin in this group of patients, the investigators have raised the need to develop a prospective observational study; describing a PK / PD model of amikacin in newborns with suspected sepsis.

DETAILED DESCRIPTION:
Three blood samples will be taken from each of the 138 participants. As a standard of care, a sample will always be taken at 0.5h (Cmax) after the first dose and a sample before the second dose, which can be at 24h, 36h, or 48h as per physician indication. The third sample will be collected according to what has been assigned by a block randomization method, in one of the following moments: 1, 2, 4, 8, 12 or 18 hours after the administration of the first dose of Amikacin.

The methods used to analyze the samples will be: Particle Enhanced Turbidimetric Immunoassay (PETIA), Architect C8000; and Homogeneous Microparticle Immunoassay in Solution (KIMS), Roche systems. The determination of the susceptibility and minimum Inhibitory Concentration (MIC) will be carried out by the laboratories of each hospital by agar dilution method.

PK/PD profile of amikacin will be evaluated with NONMEM (non-linear mixed effects modelling) software for the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Receive at least one dose of Amikacin
* Be at least three days old (72 hours)

Exclusion Criteria:

* Receive the first dose of Amikacin in a healthcare center other than those included in the research
* Patient on renal replacement therapy

Ages: 3 Days to 1 Month | Sex: All
Age Groups: Child
Study Population: Patients admitted to neonatal intensive care units of two hospitals of high-complexity in Chile
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
Volume of Distribution (L/Kg) of Amikacin | first dose amikacin (1 day)
  The mean population parameter and their interindividual variability in neonates with suspected sepsis
Clearance (L/h) of Amikacin | first dose amikacin (1 day)
  The mean population parameter and their interindividual variability in neonates with suspected sepsis
PK/PD targets of amikacin | first dose amikacin (1 day)
  Peak Plasma Concentration (Cmax) over 8 fold Minimum Inhibitory Concentration (MIC) or Cmax: 24-35 mg/L

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas F Severino, PharmD, Principal Investigator — Facultad de Medicina. Pontificia Universidad Católica de Chile
Locations (1):
- Hospital Clínico UC-Christus, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lingvall M, Reith D, Broadbent R. The effect of sepsis upon gentamicin pharmacokinetics in neonates. Br J Clin Pharmacol. 2005 Jan;59(1):54-61. doi: 10.1111/j.1365-2125.2005.02260.x. PMID 15606440
- [Background] Sherwin CM, Svahn S, Van der Linden A, Broadbent RS, Medlicott NJ, Reith DM. Individualised dosing of amikacin in neonates: a pharmacokinetic/pharmacodynamic analysis. Eur J Clin Pharmacol. 2009 Jul;65(7):705-13. doi: 10.1007/s00228-009-0637-4. Epub 2009 Mar 21. PMID 19305985